CLINICAL TRIAL: NCT01883856
Title: Comparison of Silicone and Porous Plate Ahmed Glaucoma Valves
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter Netland, MD (Other)
Collaborators: New World Medical, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Peter Netland, MD, Chair, Department of Ophthalmology, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16051
Record Dates: First submitted 2013-06-18; First posted 2013-06-21 (Estimated); Results first posted 2020-09-18 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Glaucoma
Keywords: Refractory Glaucoma; Intractable Glaucoma; Primary Open Angle Glaucoma; Neovascular Glaucoma
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Glaucoma, Neovascular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Silicone Plate Ahmed Glaucoma Valve (Active Comparator): Silicone plate Ahmed Glaucoma Valve
  Interventions: Device: Silicone plate Ahmed Glaucoma Valve (Model FP7)
- Porous Plate Ahmed Glaucoma Valve (Experimental): Porous Plate Ahmed Glaucoma Valve
  Interventions: Device: Porous Plate Ahmed Glaucoma Valve (Model M4)

INTERVENTIONS:
Device: Silicone plate Ahmed Glaucoma Valve (Model FP7) — This intervention is conducted as a surgical intervention.
  Arms: Silicone Plate Ahmed Glaucoma Valve
Device: Porous Plate Ahmed Glaucoma Valve (Model M4) — This intervention is conducted as a surgical intervention.
  Arms: Porous Plate Ahmed Glaucoma Valve

SUMMARY:
The purpose of this study is to evaluate and compare the clinical outcomes after implantation of the porous plate (polyethylene) (Model M4) Ahmed Glaucoma Valve with the silicone plate Ahmed Glaucoma Valve (Model FP7) in participants with refractory glaucoma.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate and compare the clinical outcomes after implantation of the porous plate (polyethylene) (Model M4) Ahmed Glaucoma Valve with the silicone plate Ahmed Glaucoma Valve (Model FP7) in participants with refractory glaucoma. Participation will last for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any race ≥ 18 years and ≤ 80 years of age.
* Diagnosis of intractable glaucoma in the study eye, with the exception of silicone oil endotamponade induced glaucoma, which has not responded to conventional medical and surgical therapy.
* Elevated intraocular pressure > 21 mmHg in the study eye. Two consecutive measurements using Goldmann Applanation Tonometry will be obtained and the mean of those two measurements will be considered the subject's baseline intraocular pressure.
* Subject is a candidate for surgery in the study eye with a glaucoma drainage device.
* Subject is willing and able to sign the informed consent.

Exclusion Criteria:

* Diagnosis of silicone oil endotamponade induced glaucoma in the study eye.
* History of prior drainage implant surgery in the study eye.
* History of cyclophotocoagulation of the study eye.
* Pregnancy.
* Prisoner.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-02; Primary Completion 2017-09-10 (Actual); Study Completion 2018-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Netland, MD, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Described in study results - https://pubmed.ncbi.nlm.nih.gov/32765127/

REFERENCES:
- [Result] Roa TM, Netland PA, Costa VP, Sarkisian SR Jr, Al-Aswad LA, Moster MR, Ahmed IIK. Comparison of Silicone- and Porous-Plate Ahmed Glaucoma Valves. Med Devices (Auckl). 2020 Jul 16;13:213-221. doi: 10.2147/MDER.S258498. eCollection 2020. PMID 32765127
- See also: Study results indexed on Pub Med — https://pubmed.ncbi.nlm.nih.gov/32765127/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Silicone Plate Ahmed Glaucoma Valve | Porous Plate Ahmed Glaucoma Valve
Started | 26 | 26
Completed | 26 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Silicone Plate Ahmed Glaucoma Valve | Porous Plate Ahmed Glaucoma Valve | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (11.2) | 67.0 (10.1) | 67.3 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 13 | 18 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: African American | 8 | 9 | 17
  Ethnicity: Asian | 2 | 0 | 2
  Ethnicity: Caucasian | 14 | 14 | 28
  Ethnicity: Hispanic | 1 | 3 | 4
  Ethnicity: Mixed Race | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 21 | 38
  Canada | 2 | 0 | 2
  Brazil | 7 | 5 | 12
Pre-operative intraocular pressure [Mean (Standard Deviation); unit: mmHg] | 29.91 (6.55) | 33.79 (10.54) | 31.85 (8.55)

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Pressure
Description: The primary endpoint is the mean intraocular pressure in the porous plate group as compared to the silicone plate group.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Silicone Plate Ahmed Glaucoma Valve | Porous Plate Ahmed Glaucoma Valve
Number analyzed (Participants) | 26 | 26
mmHg | 13.60 (4.69) | 17.94 (10.95)

2. Secondary Outcome: Anti-Glaucoma Medications
Description: The mean number of anti-glaucoma medications in the porous plate group as compared to the silicone plate group at 12 months.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: glaucoma medications
Arm/Group | Silicone Plate Ahmed Glaucoma Valve | Porous Plate Ahmed Glaucoma Valve
Number analyzed (Participants) | 26 | 26
glaucoma medications | 1.64 (1.40) | 1.89 (1.54)

3. Secondary Outcome: Surgical Success
Description: Surgical success in the porous plate group as compared to the silicone plate group at 12 months. Surgical success was defined as intraocular pressure of ≤5 mmHg or ≥21 mmHg (with or without glaucoma medications), with no loss of light perception, and no additional glaucoma procedures.
Time Frame: 12 months
Measure: Number; unit: surgical success
Arm/Group | Silicone Plate Ahmed Glaucoma Valve | Porous Plate Ahmed Glaucoma Valve
Number analyzed (Participants) | 26 | 26
surgical success | 23 | 14

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Silicone Plate Ahmed Glaucoma Valve | Porous Plate Ahmed Glaucoma Valve
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 13/26 | 15/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silicone Plate Ahmed Glaucoma Valve (N=26) | Porous Plate Ahmed Glaucoma Valve (N=26)
Hypertensive phase (Eye disorders) | 13 (13) | 15 (15) — Hypertensive phase was defined as intraocular pressure more than 21 mmHg during the first three months postoperatively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-25): https://cdn.clinicaltrials.gov/large-docs/56/NCT01883856/Prot_SAP_000.pdf